CLINICAL TRIAL: NCT04012840
Title: Determinant of the Risk of the Becoming Frail in the Non-dependent Elederly
Acronym: DEPART
Status: Recruiting | Type: Observational
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A00254-51
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Risk of Frailty in Elderly
Keywords: Frailty; Fried's criteria; Rockwood's criteria; Loss of autonomy,; elderly
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
As an active and healthy ageing, "Successful Ageing" is a societal challenge for all countries members according to the European Commission. This study is intended to contribute to increase healthy, active and non-dependent lifetime. To this end the main goal is to highlight clinical and biological frailty determinants in elderly with potential weaknesses.

DETAILED DESCRIPTION:
Detailed Description:

Definition: Extended description of the protocol, including more technical information (as compared to the Brief Summary) if desired. Do not include the entire protocol; do not duplicate information recorded in other data elements, such as eligibility criteria or outcome measures.

Example:

Sudden out-of-hospital cardiac arrest (OOH-CA) remains a significant cause of death, in spite of recent declines in overall mortality from cardiovascular disease. Existing methods of emergency resuscitation are inadequate due to time delays inherent in the transport of a trained responder with defibrillation capabilities to the side of the OOH-CA victim. Existing Emergency Medical Services (EMS) systems typically combine paramedic Emergency Medical Technician (EMT) services with some level of community involvement, such as bystander cardiopulmonary resuscitation (CPR) training. Some communities include automated external defibrillators (AEDs) at isolated sites or in mobile police or fire vehicles. A comprehensive, integrated community approach to treatment with AEDs would have community units served by these volunteer non-medical responders who can quickly identify and treat a patient with OOH-CA. Such an approach is termed Public Access Defibrillation (PAD). Healthy, active and non-dependent lifetime during ageing is a societal challenge for European Union. One of the worst consequences of ageing is the loss of autonomy which may be preceded by a mid-state between good and pathological ageing. This mid-state is called "frailty syndrome" and cause a lot of hospitalizations (Morley et al., 2013). This statement is potentially reversible if early procedures mixing geriatric interventions based on standardised geriatric evaluation and general practitioners cooperation are established (Haute Autorité de Santé, 2013). The main studied interventions are physical training, cognitive stimulation and nutritional actions (Bibas et al., 2014; Clegg et al., 2013). Frailty syndrome is a geriatric syndrome emphasizes by the homeostatic reserves drop which induces a stress response failure and expose the person to a wrong medical prognosis (Clegg et al., 2013; Rodriguez-Manas et al., 2013; Rolland et al., 2011). Its clinical expression is modulated by comorbidities and psychological, social, economic and behavioural factors. Thus, frailty syndrome is a mortality risk and pejorative events factor, especially those of loss of autonomy, falls, hospitalizations and institutionalization in a 1 to 3 years delay. So, the main goal is to highlight clinical and biological frailty determinants in elderly with potential weaknesses. If there is no strict frailty definition, two frailty criteria types are officially used :

1. Fried's criteria are the more commonly used criteria to diagnose frailty (Fried et al., 2001):

   * Involuntary weight loss > 4.5 kg in one year,
   * A feeling of exhaustion,
   * Low muscle strength (handgrip <20% norm for age, sex and self- bmi),
   * Low physical activity (<383 kcal/week spent for men, <270kcal/week for women)
   * Low walking speed (<0.8m/s). According to the number of Fried's criteria, subjects are considered frail (≥ 3 criteria), pre-frail (1-2 criteria) or robust (0 criterion).
2. Rockwood (Rockwood et al., 2005) or Winograd's criteria (Winograd et al., 1988) based on the mix of medical and social factors also known as "multidomain frailty" incorporate additional pattern of comorbidities (70 parameters in Rockwood's criteria) and geriatric syndromes (confusion, dementia, bed sores, falls, malnourishment…) which actually are too general and leading to detect patients too late.

To diagnose and evaluate this frailty a global geriatric evaluation based on the multidimensional comprehensive geriatric assessment (Haute Autorité de Santé, 2013) must be led, which is a long process specifically realized in geriatrics. Due to several limits in both Fried' and Rockwood's criterion. In Fried's model the slow of walking speed is hard to evaluate, the exhaustion of the patient can depend on a previous psychological state (Drey et al., 2011), also the measure of muscle strength which requires a dynamometer is not always achievable for example. Likewise, in Rockwood's criteria the whole 70 variables are too long to list, even under its short form which includes 30 variables.

Thus, since there is no easy-to-use consensual tool, the real frailty in elderly is nowadays rarely detected. Yet it remains essential to identify the mains biological or clinical factors which will forecast the loss of autonomy. The highlighting of those factors would allow an earlier screening in order to propose several interventions to delay the loss of autonomy.

Non interventional and prospective study in which recruitment and frailty evaluation will be realized in a special geriatric ward (medical examination in day hospital and preventive center). This study bases its choice of patient on the results of a 6 questions survey (from the Gérontopôle of Toulouse) about frailty.

* The main objective is to highlight the clinical and biological determinants of loss of autonomy in non-dependent and potentially frail elderly.
* Secondaries objectives are to highlight the clinical and biological determinants of loss of autonomy in non-dependent and potentially frail elderly by testing :

  * Cognitive disorders;
  * Risk of falls;
  * Malnourishment;
  * Depression;
  * New illnesses appearances;
  * Unscheduled hospitalizations;
  * Mortality;
  * Institutionalization;
* Evaluate the impact of the geriatrician subjective impression on the loss of autonomy.

People will be recruited among patients whose consult in prevention centers and day hospitals in Île-de-France :

* 9 geriatric centers
* 2000 patients will be included over 36 months
* Approximatively 7 patients per week in each center
* Inclusions will take place for 3 years
* A following up call every 6 months for 3 years

ELIGIBILITY:
Inclusion criteria :

* Age ≥ 70 years old
* Patient with frailty risks according to a survey recommended by HAS (Gérontopôle of Toulouse)
* ADL≥5
* Agreeing to take part in a geriatric assessment in a prevention center or in a Day hospital in Île-de-France
* Agreeing to be followed by phone every 6 months for 3 years
* Eligible to a social security system

Exclusion criteria :

* A stated loss of autonomy
* Individual under guardianship, curatorship, judicial supervision

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: : +70 years old elderly with a potential frailty whose accept to participate to a geriatric assessment in a prevention center or in a day hospital and to be followed bwith phone calls every 6 months for 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-06-26 (Actual); Primary Completion 2030-06-25 (Estimated); Study Completion 2030-12-25 (Estimated)

PRIMARY OUTCOMES:
Loss of 1 or more point in activities of daily living (ADL) score which assert a loss of autonomy - Loss of 1 or more point in instrumental activities of daily living (IADL) score which assert a loss of autonomy During the monitoring, those evaluatio | 3 years

SECONDARY OUTCOMES:
Assessment of ccurrence of cognitive disorders according Mini Mental State Examination (MMSE) | 3 years
Occurrence of drivers of risk of falls : search for orthostatic hypotension (occurrence or missing), leg stance, tandem station, SPPB, TUG, grip force. | 3 years
Constated malnourishment according Mini Nutritional Assessment MNA short form | 3 years
Occurrence of a depression according Mini Geriatric Depression Scale "mini GDS" ≥ 1 | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hanon, MD PhD, Study Chair — Geriatrci Department, Broca Hospital
Locations (1):
- Geriatric Department, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No